CLINICAL TRIAL: NCT05499910
Title: Training in Neuro Strengths-Based Approach to Autism
Brief Title: Neuro Strengths-Based Approach to Autism
Acronym: NSBAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baio Enterprises (Other)
Collaborators: Baio Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015835
Record Dates: First submitted 2022-07-18; First posted 2022-08-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSBAA (Experimental): The Neuro Strengths-Base Approach to Autism is an approach developed from various research on how the autistic brain works, the approaches that work best to motivate autistic individuals, and how others can understand as well as support behaviors that may occur with autistic individuals.
  Interventions: Behavioral: NSBAA

INTERVENTIONS:
Behavioral: NSBAA — The Neuro Strengths-Based Approach to Autism is an approach that teaches people how the autistic brain works and the best practices for providing intervention.

SUMMARY:
The Neuro-Strength-Based Approach to Autism (NSBAA) attempts to translate what research has discovered about the autistic brain into terms that autistics, and those involved with autistics, can understand. It is not intended to be a new approach to intervention but hopefully a unifying approach to understanding autism that all therapists, educators, clinicians, and parents can use when working with autistic individuals. It was developed by an autistic occupational therapist, based on her lifetime obsession of learning everything she could about how typical brains work, and, following her diagnosis, how the autistic brain works. Being on the autism spectrum herself and having worked with, and interacted with, autistic individuals of all ages and abilities in school, clinical, and personal settings, the author attempts to explain the autistic brain from both the scientific as well as autistic perspectives.

ELIGIBILITY:
Inclusion Criteria:

* 5-20 SLPs / OTR/Ls, regardless of nationality
* working in a clinical, home or school setting with less than 25 years of experience
* at least 2 years of experience working with autistic clients

Exclusion Criteria:

* Minors
* adults unable to consent
* undocumented individuals
* prisoners,
* uncertified therapists
* therapists from Baio Enterprises.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Measurable change in the participant's satisfaction with their ability to write neuro-strength-based goals | After 16 hours of training
  Participants will show a significant increase (50% or higher) in their ratings on the NSBSA Satisfaction With Writing and Implementing Goals For Autistic Clients given to them pre-training, 3 months post-training, and 6 months post-training. They will rate their satisfaction with 28 elements included in the NSBSA Training Modules using a rating scale of 1-5, with 1 being very dissatisfied and 5 being very satisfied. The highest possible score is 140 and the lowest is 28.
Measurable change in participants' knowledge of the clinical reasoning for the goals they write | After 16 hours of training
  Participants will show a significant increase (50% or higher) in the number of goal components they are able to include in their goal, with a maximum of 8, and the number of questions that challenge their reasoning for what they include, with a maximum of 23, in the goals they submit using the Pre- and Post-Training Goal Writing Forms. The highest possible score is 31 if they complete all components and answer all questions. The lowest possible score is 0.

SECONDARY OUTCOMES:
Measurable change in the completeness of the goals: | After 16 hours of training
  Participants will show a significant increase (50% or higher) in the score they receive on the Post-Training Goal Writing Form compared to the Pre-Training Goal Writing Form, using the Pre-and Post-Training Scoring for Goal Writing Form, with the highest possible score being +32 and the lowest score being -16 with an average score of 0.

CONTACTS AND LOCATIONS:
Overall Officials: Blair Braden, PhD, Principal Investigator — Arizona State University
Locations (1):
- Staci L Neustadt, Littleton, Colorado, United States

REFERENCES:
- [Background] Wolff, Michael. (2018). The Complexity of Autism Spectrum Disorders
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders. Washington DC: American Psychiatric Association; 2013. 646
- [Background] Wozniak RH, Leezenbaum NB, Northrup JB, West KL, Iverson JM. The development of autism spectrum disorders: variability and causal complexity. Wiley Interdiscip Rev Cogn Sci. 2017 Jan;8(1-2):10.1002/wcs.1426. doi: 10.1002/wcs.1426. Epub 2016 Dec 1. PMID 27906524
- [Background] Ha S, Sohn IJ, Kim N, Sim HJ, Cheon KA. Characteristics of Brains in Autism Spectrum Disorder: Structure, Function and Connectivity across the Lifespan. Exp Neurobiol. 2015 Dec;24(4):273-84. doi: 10.5607/en.2015.24.4.273. Epub 2015 Dec 16. PMID 26713076
- [Background] Riosa, Priscilla & Chan, Victoria & Maughan, Andrea & Stables, Victoria & Albaum, Carly & Weiss, Jonathan. (2017). Remediating Deficits or Increasing Strengths in Autism Spectrum Disorder Research: a Content Analysis. Advances in Neurodevelopmental Disorders. 1. 10.1007/s41252-017-0027-3.
- [Background] Urbanowicz A, Nicolaidis C, den Houting J, Shore SM, Gaudion K, Girdler S, Savarese RJ. An Expert Discussion on Strengths-Based Approaches in Autism. Autism Adulthood. 2019 Jun 1;1(2):82-89. doi: 10.1089/aut.2019.29002.aju. Epub 2019 Apr 13. No abstract available. PMID 36601531
- [Background] Donaldson A, Krejcha K, McMillin A. A Strengths-Based Approach to Autism: Neurodiversity and Partnering With the Autism Community. Perspectives of the ASHA Special Interest Groups (2017) 2(1) 56-68
- [Background] Patten Koenig K. A strength-based frame of reference for autistic individuals. Frames of reference for pediatric occupational therapy (4th edition) (2019)
- [Background] Patten Koenig K. Authentic Strength-Based Practice: Can Neurotypical Professionals Make a Paradigm Shift? Autism Spectrum News (2020) (Winter)
- [Background] Leadbitter K, Buckle KL, Ellis C, Dekker M. Autistic Self-Advocacy and the Neurodiversity Movement: Implications for Autism Early Intervention Research and Practice. Front Psychol. 2021 Apr 12;12:635690. doi: 10.3389/fpsyg.2021.635690. eCollection 2021. PMID 33912110